CLINICAL TRIAL: NCT02657902
Title: Does an Additional Antirotation U-Blade (RC) Lagscrew Improve Treatment of AO/OTA (Orthopaedic Trauma Association) 31 A1-3 Classified Fractures With Gamma 3 Nail?
Brief Title: Does an Additional Antirotation U-Blade (RC) Lagscrew Improve Treatment of AO/OTA (Orthopaedic Trauma Association) 31 A1-3 Fractures With Gamma 3 Nail?
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Julian Joestl, MD, Medical University of Vienna
Other Study IDs: 1960/2015
Record Dates: First submitted 2016-01-08; First posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Gamma 3 Nail: Fractures that were treated with a Gamma 3 nail
  Interventions: Procedure: Fractures were treated with a Gamma 3 intramedullary nail
- Gamma 3 Nail + U-Blade: Fractures that were treated with a Gamma 3 nail and additional with antirotation U-blade lag screws.
  Interventions: Procedure: Fractures were treated with a Gamma 3 intramedullary nail + U-Blade

INTERVENTIONS:
Procedure: Fractures were treated with a Gamma 3 intramedullary nail
  Groups: Gamma 3 Nail
Procedure: Fractures were treated with a Gamma 3 intramedullary nail + U-Blade
  Groups: Gamma 3 Nail + U-Blade

SUMMARY:
The purpose was to evaluate whether the additional use of the Gamma3 ® RC Lag Screw is associated with a reduced cutout rate in patients with OTA/AO 31A1-3 inter-trochanteric fractures.

ELIGIBILITY:
Inclusion Criteria:

* OTA/AO 31A1-3 fractures treated with Gamma 3® Nail (Stryker Trauma Germany) and either with standard lagscrews or with the Gamma3 ® RC Lag Screw (Stryker Trauma Germany)

Exclusion Criteria:

* Patients with pathological fractures
* Patients treated with a long gamma nail were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with OTA/AO 31A1-3 fractures treated with Gamma 3® Nail (Stryker Trauma Germany) and either with standard lagscrews or with the Gamma3 ® RC Lag Screw (Stryker Trauma Germany)
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2009-01; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Cutout rate | 3 months after intervention
  Differences in the Cutout rate of the femoral head screw with/without U-Blade antirational screw

SECONDARY OUTCOMES:
Mobility | 3 months after intervention
  Mobility of the patients 3 months after intervention measured with the Parker mobility score